CLINICAL TRIAL: NCT00213798
Title: Detection of Plasma DNA by Allelotyping in Non Small Cell and Small Cell Lung Cancer Patients. Evolution During Treatment and Follow-up.
Brief Title: Detection of Plasma DNA in Non Small Cell and Small Cell Lung Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2731
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Carcinoma; Small Cell Lung Cancer
Keywords: Lung cancer; plasma DNA; allelotyping; follow-up; Prospective Study; Non-Small Cell Lung Cancer; Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Lung Neoplasms

INTERVENTIONS:
Procedure: Biopsy samples

SUMMARY:
The majority of lung cancer patients have a tumor-derived genetic alteration in circulating plasma DNA that could be exploited as a diagnostic tool. The aim of this study is to evaluate if plasma DNA can be used as a valuable non invasive test to monitor disease progression without assessing the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Presence of lung tumor to use fiberoscopy or surgical intervention for diagnosis.
* No lung instability.
* Individuals give all informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2003-12; Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michèle BEAU-FALLER, MD, Principal Investigator — Service de Pneumologie, Hôpital de Hautepierre
Locations (4):
- France (4):
  - Service de Pneumologie, Hôpital Lyautey, Strasbourg
  - Service de Chirurgie Thoracique, Hôpital Civil, Strasbourg
  - Service de Pneumologie, Hôpital Civil, Strasbourg
  - Service de Pneumologie, Hôpital de Hautepierre, Strasbourg

REFERENCES:
- [Result] Beau-Faller M, Gaub MP, Schneider A, Ducrocq X, Massard G, Gasser B, Chenard MP, Kessler R, Anker P, Stroun M, Weitzenblum E, Pauli G, Wihlm JM, Quoix E, Oudet P. Plasma DNA microsatellite panel as sensitive and tumor-specific marker in lung cancer patients. Int J Cancer. 2003 Jun 20;105(3):361-70. doi: 10.1002/ijc.11079. PMID 12704670